CLINICAL TRIAL: NCT02127593
Title: A Single-Dose, Open-Label, Randomized, 2-Way Crossover Pivotal Study to Assess the Bioequivalence of NGM/EE Tablets Manufactured at 2 Different Facilities
Brief Title: A Bioequivalence Study of Norgestimate /Ethinyl Estradiol (NGM/EE) Tablets Manufactured at 2 Different Facilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR104172; 10131CON1001 (Other: Janssen Research & Development, LLC); 2014-000983-16 (EudraCT Number)
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Norgestimate; Ethinyl estradiol; Norgestrel; Norelgestromin; Ortho cyclen; Phase 1; Healthy Women
MeSH Terms: interventions — norgestimate; Ethinyl Estradiol; cyclen; Moxifloxacin; norgestimate, ethinyl estradiol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First NGM/EE (Wet Process), then NGM/EE (Dry Process) (Experimental): Participants will receive 1 tablet (formulated by wet process) containing norgestimate 250 microgram (mcg) and ethinyl estradiol 35 mcg, orally on Day 1 of Period 1, followed by 1 tablet (formulated by dry process) containing norgestimate 250 mcg and ethinyl estradiol 35 mcg, orally on Day 1 of Period 2, wherein Period 1 and Period 2 are separated by a wash out period of at least 10 days.
  Interventions: Drug: Norgestimate /Ethinyl estradiol tablets (NGM/EE) (Wet Process); Drug: Norgestimate /Ethinyl estradiol tablets (NGM/EE) (Dry Process)
- First NGM/EE (Dry Process), then NGM/EE (Wet Process) (Experimental): Participants will receive 1 tablet (formulated by dry process) containing norgestimate 250 mcg and ethinyl estradiol 35 mcg, orally on Day 1 of Period 1, followed by 1 tablet (formulated by wet process) containing norgestimate 250 mcg and ethinyl estradiol 35 mcg, orally on Day 1 of Period 2, wherein Period 1 and Period 2 are separated by a wash out period of at least 10 days.
  Interventions: Drug: Norgestimate /Ethinyl estradiol tablets (NGM/EE) (Wet Process); Drug: Norgestimate /Ethinyl estradiol tablets (NGM/EE) (Dry Process)

INTERVENTIONS:
Drug: Norgestimate /Ethinyl estradiol tablets (NGM/EE) (Wet Process) — Norgestimate /Ethinyl estradiol tablets (NGM/EE) containing norgestimate 250 mcg and ethinyl estradiol 35 mcg, formulated by wet process will be orally administered on Day 1 of Period 1 or Period 2.
  Other Names: Cyclen; Tri Cyclen; Cilest; Tri-Cilest
Drug: Norgestimate /Ethinyl estradiol tablets (NGM/EE) (Dry Process) — Norgestimate /Ethinyl estradiol tablets (NGM/EE) containing norgestimate 250 mcg and ethinyl estradiol 35 mcg, formulated by dry process will be orally administered on Day 1 of Period 1 or Period 2.
  Other Names: Ortho Cyclen; Ortho Tri Cyclen

SUMMARY:
The purpose of this study is to establish the bioequivalence of the hormones norgestimate, norelgestromin, and ethinyl estradiol in norgestimate/ethinyl estradiol (NGM/EE) tablets, formulated by wet process compared with the same hormones in NGM/EE tablets, formulated by dry process, in healthy women.

DETAILED DESCRIPTION:
This is a Phase 1, single-dose, open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), randomized (the study medication is assigned by chance), single-center and a 2-way crossover (method used to switch participants from one study group to another in a clinical trial) study in healthy women. The study consists of 3 parts: Screening phase, Treatment phase and end-of-study or withdrawal. Treatment periods will be separated by a wash out period of at least 10 days. The duration of participation in the study for an individual participant will be approximately 7 weeks. All participants will be randomly assigned in a 1:1 ratio to 1 of 2 possible treatment sequences and receive both of the following treatments: 1 oral tablet formulated by wet process or dry process, whereas each tablet contains norgestimate 250 microgram (mcg) and ethinyl estradiol 35 mcg. The primary endpoint of the study will be assessment of pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be either surgically sterile or of child-bearing potential and be practicing an effective non-hormonal method of birth control (for example, copper intrauterine device, double-barrier method, male partner sterilization) before entry and throughout the study
* If a woman of child-bearing potential, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative urine pregnancy test on Day -1 of the each treatment period
* Participants must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after the last dose
* Body mass index (BMI: weight [kilogram {kg}]/height^2 [meter {m}]^2) between 18.5 and 30 kg/m^2 (inclusive), and body weight not less than 50 kilogram (kg) or higher than 90 kg (198 pounds)
* Participant must be a non-smoker

Exclusion Criteria:

* Participants have a levonorgestrel implant (for example, Norplant) in place or removed within the 30 days before admission to the study site
* Contraindications to combined hormonal contraceptives
* Participants who received medroxyprogesterone injection (for example, Depo Provera) within 6 months of admission to the study
* Use of any other hormonal contraceptive within 30 days of admission to the study site
* Participants with abnormal papanicolaou (Pap) smear or CytoRich test

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (C[max]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  The C(max) is the maximum serum concentration which will be observed at the defined time points.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  The AUC (last) is the area under the plasma concentration-time curve from time zero time of the last quantifiable concentration C(last), and C(last) is the last observed quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  The AUC (infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Time to Reach the Maximum Plasma Concentration (T[max]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  The T[max] is time to reach the observed maximum plasma concentration.
Percentage of AUC(0-infinity) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  Percentage of AUC(0-infinity) is calculated as (AUC[0-infinity] minus AUC[0-last] divided by AUC[0-infinity]) multiplied by 100.
Elimination Half-life Period (t1/2) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  Elimination half-life associated with the terminal slope (lambda[z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda (z).
Terminal slope (Lambda [z]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  Terminal slope is defined by first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Coefficient of Determination (r^2) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  The coefficient of determination is a goodness of fit statistic that gives the proportion of the variance of one variable that is predictable from the other variable.
Adjusted Coefficient of Determination (r^2 adj.) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 72 hours after study drug administration on Day 1 of Period 1 and Period 2
  The coefficient of determination adjusted (r^2 adj.) for the number of points used in the estimation of lambda[z].

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (1):
- Groningen, Netherlands